CLINICAL TRIAL: NCT00664287
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 12-Week Study to Evaluate the Efficacy and Safety of Extended Release (ER) Niacin/Laropiprant When Added to Ongoing Lipid-Modifying Therapy in Dyslipidemic Patients Deemed Appropriate for Further Lipid Modification.
Brief Title: Extended Release (ER) Niacin/Laropiprant Add on Study (0524A-082)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-082; 2008_504
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Experimental): Patients will remain on existing lipid-modifying therapy throughout the study. Group 1: Patients will receive ER niacin/laropiprant 1 g/20 mg daily. After 4 weeks, ER niacin/laropiprant will be increased to 2 g/40 mg for remainder of study.
  Interventions: Drug: niacin (+) laropiprant
- Group 2 (Placebo Comparator): Patients will remain on existing lipid-modifying therapy throughout the study. Group 2: Patients will receive 1 placebo tablet daily. After 4 weeks, patients will be advanced to 2 placebo tablets for remainder of the study.
  Interventions: Drug: placebo (unspecified)

INTERVENTIONS:
Drug: niacin (+) laropiprant — Group 1: Patients will receive ER niacin/laropiprant 1 g/20 mg daily. After 4 weeks, ER niacin/laropiprant will be increased to 2 g/40 mg for remainder of study.
  Other Names: MK0524A
  Arms: Group 1
Drug: placebo (unspecified) — Group 2: Patients will receive 1 placebo tablet daily. After 4 weeks, patients will be advanced to 2 placebo tablets for remainder of the study.
  Arms: Group 2

SUMMARY:
The purpose of this study is to test the effect of MK0524A (niacin (+) laropiprant) on lowering bad cholesterol and raising good cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older and on a stable dose of lipid therapy

Exclusion Criteria:

* Patients lipid level is outside the recommended range
* Patients that are HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Lipid modification results of MK0524A (niacin (+) laropiprant) compared to placebo on LDL-C throughout the study and at 17 weeks. | 3 months

SECONDARY OUTCOMES:
Lipid modification results of MK0524A (niacin (+) laropiprant) on blood lipids such as LDL-C, HDL-C, triglycerides, etc., throughout the study and at 17 weeks. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC